CLINICAL TRIAL: NCT00076089
Title: Effect of Roflumilast on Exacerbation Rate in Patients With Chronic Obstructive Pulmonary Disease. A 52-week, Multicenter, Double-blind Study With 500 mcg Roflumilast Once Daily Versus Placebo.
Brief Title: OPUS Study: Effect of Roflumilast on Exacerbation Rate in Patients With Chronic Obstructive Pulmonary Disease (BY217/M2-111)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-111
Record Dates: First submitted 2004-01-13; First posted 2004-01-15 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Roflumilast; Chronic obstructive pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The purpose of this study is to determine whether roflumilast is effective in the treatment of exacerbations in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Main Inclusion Criteria:

* FEV1/FVC ratio (post-bronchodilator) ≤70%
* FEV1 (post-bronchodilator) ≤50% of predicted
* Current smoker or ex-smoker
* Clinically stable COPD indicated by no exacerbation and no change in COPD treatment of within 4 weeks prior to baseline
* Availability of chest x-ray dated a maximum of 6 months prior to study baseline or a willingness to have a chest x-ray performed at baseline

Main Exclusion Criteria:

* COPD exacerbation indicated by a treatment with systemic glucocorticoids not stopped 4 weeks prior to baseline
* Lower respiratory tract infection not resolved 4 weeks prior to baseline
* Diagnosis of asthma and/or other relevant lung disease
* Known alpha-1-antitrypsin deficiency
* Need for long-term oxygen therapy defined as ≥16 hours/day

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2003-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
change in FEV1 from baseline during the treatment period; number of COPD exacerbations.

SECONDARY OUTCOMES:
pulmonary function variables
number of COPD exacerbations of different type and various subgroups
quality of life variables
patient diary variables
time to study withdrawal
safety.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (40):
- United States (35):
  - ALTANA Pharma, Cities in Alabama, Alabama
  - ALTANA Pharma, Cities in Arizona, Arizona
  - ALTANA Pharma, Cities in Arkansas, Arkansas
  - ALTANA Pharma, Cities in California, California
  - ALTANA Pharma, Cities in Colorado, Colorado
  - ALTANA Pharma, Cities in Connecticut, Connecticut
  - ALTANA Pharma, Cities in Florida, Florida
  - ALTANA Pharma, Cities in Georgia, Georgia
  - ALTANA Pharma, Cities in Illionois, Illinois
  - ALTANA Pharma, Cities in Iowa, Iowa
  - ALTANA Pharma, Cities in Kentucky, Kentucky
  - ALTANA Pharma, Cities in Louisiana, Louisiana
  - ALTANA Pharma, Cities in Massachusetts, Massachusetts
  - ALTANA Pharma, Cities in Minnesota, Minnesota
  - ALTANA Pharma, Cities in Missouri, Missouri
  - ALTANA Pharma, Cities in Montana, Montana
  - ALTANA Pharma, Cities in Nebraska, Nebraska
  - ALTANA Pharma, Cities in Nevada, Nevada
  - ALTANA Pharma, Cities in New Hampshire, New Hampshire
  - ALTANA Pharma, Cities in New Jersey, New Jersey
  - ALTANA Pharma, Cities in New York, New York
  - ALTANA Pharma, Cities in North Carolina, North Carolina
  - ALTANA Pharma, Cities in Ohio, Ohio
  - ALTANA Pharma, Cities in Oklahoma, Oklahoma
  - ALTANA Pharma, Cities in Oregon, Oregon
  - ALTANA Pharma, Cities in Pennsylvania, Pennsylvania
  - ALTANA Pharma, Cities in Rhode Island, Rhode Island
  - ALTANA Pharma, Cities in South Carolina, South Carolina
  - ALTANA Pharma, Cities in Tennessee, Tennessee
  - ALTANA Pharma, Cities in Texas, Texas
  - ALTANA Pharma, Cities in Utah, Utah
  - ALTANA Pharma, Cities in Vermont, Vermont
  - ALTANA Pharma, Cities in Virginia, Virginia
  - ALTANA Pharma, Cities in West Virginia, West Virginia
  - ALTANA Pharma, Cities in Wisconsin, Wisconsin
- ALTANA Pharma, Cities in Canada, Canada
- ALTANA Pharma, Cities in France, France
- ALTANA Pharma, Cities in Germany, Germany
- ALTANA Pharma, Cities in Poland, Poland
- ALTANA Pharma, Cities in South Africa, South Africa

REFERENCES:
- [Derived] Facius A, Krause A, Claret L, Bruno R, Lahu G. Modeling and Simulation of Pivotal Clinical Trials Using Linked Models for Multiple Endpoints in Chronic Obstructive Pulmonary Disease With Roflumilast. J Clin Pharmacol. 2017 Aug;57(8):1042-1052. doi: 10.1002/jcph.885. Epub 2017 Apr 17. PMID 28419462
- [Derived] Rennard SI, Calverley PM, Goehring UM, Bredenbroker D, Martinez FJ. Reduction of exacerbations by the PDE4 inhibitor roflumilast--the importance of defining different subsets of patients with COPD. Respir Res. 2011 Jan 27;12(1):18. doi: 10.1186/1465-9921-12-18. PMID 21272339
- See also: BY217-M2-111-RDS-2008-12-23.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4477&filename=BY217-M2-111-RDS-2008-12-23.pdf